CLINICAL TRIAL: NCT06638060
Title: Continuous Connected Patient Care (CCPC), a Pilot Testing a Novel Device for Continuous Vitals Monitoring - Older Adults Department PHC
Status: Recruiting | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Collaborators: Excelar (Unknown); Cloud DX Inc. (Industry); Bridge Health Solutions (Unknown); Providence Healthcare (Other)
Responsible Party: Sponsor
Other Study IDs: H24-00744
Record Dates: First submitted 2024-09-16; First posted 2024-10-15 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Aging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To confirm feasibility and accessibility of the CCPC Platform (Oxymotion, Bridge Health Solutions medication adherence software, CloudDX home kit) in two different environments - 1) hospital (Acute Care for Elderly Unit) and 2) at-home .

ELIGIBILITY:
Inclusion Criteria:

* Inpatients on the Acute care of the Elderly ward.

Exclusion Criteria:

* Lack of capacity to consent to the study including moderate-severe dementia or delirium
* Unable to use (or does not have a caregiver who can help put on) study monitoring device at home
* Unable to complete (or does not have a caregiver who can help complete) study questionnaires by electronic (mobile, tablet, or computer), paper, nor phone
* Patient with known allergic reactions to any part material of the device
* People under 40kg

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The Acute Care for Elderly Unit at SPH for 40 inpatients over the age of 65.
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2025-12-21 (Estimated)

PRIMARY OUTCOMES:
Collect patient and clinicians' feedback about the CCPC Platform | From enrollment to the end of follow up at 10 days
  This will be completed via an assessment of the quantitative data on how long and how often patients use this monitoring and what were the reasons that patients took the monitors on and off.
Collect patient and clinicians' feedback about the CCPC Platform | From enrollment to the end of follow up at 10 days
  This will be completed via an assessment of the Usability Questionnaire.
Collect patient and clinicians' feedback about the CCPC Platform | From enrollment to the end of follow up at 10 days
  This will be completed by an evaluation for potential harm, e.g. anxiety questionnaire and any patient-reported adverse events.
Confirm the technical goals of the CCPC platform are met. | From enrollment to the end of follow up at 10 days
  This will be completed by ensuring clinician workflow is met, via feedback sessions (e.g. conversations, questionnaires).
Confirm the technical goals of the CCPC platform are met. | From enrollment to the end of follow up at 10 days
  This will be completed via an assessment of the data flow: does the correct patient data reach the clinicians at the right time?
Confirm the technical goals of the CCPC platform are met. | From enrollment to the end of follow up at 10 days
  This will be completed by determining if the CCPC platform provided a holistic view of each patient with vitals, medication, labs and other collected data.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Paul'sHospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No